CLINICAL TRIAL: NCT01704625
Title: Will the Use of Osteopathic Manipulative Treatments on Patients With Headache in the Emergency Department Result in Decreased Pain on 100 Point Pain Scale?
Brief Title: Will the Use of Osteopathic Manipulative Treatments Help Alleviate Headache Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Good Samaritan Hospital Medical Center, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-013
Record Dates: First submitted 2012-09-19; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Headache
Keywords: pain; headache
MeSH Terms: conditions — Headache; Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic Manipulative Treatment (Experimental): The osteopathic treatment group will have performed on them 3 standardized osteopathic manipulative treatments. If at any time the patient is unable to tolerate a treatment secondary to pain that particular study will be stopped. If the patient's nurse enters the room with medication, the study will be stopped and patient will not be included in the study. At no time will the patient's medical treatment in the emergency department be delayed to perform OMT
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Sham Osteopathic Manipulative Treatment (Sham Comparator): The sham group will receive 3 sham treatments. If at any time the patient is unable to tolerate a treatment secondary to pain that particular study will be stopped. If the patient's nurse enters the room with medication, the study will be stopped and patient will not be included in the study. At no time will the patient's medical treatment in the emergency department be delayed to perform OMT.
  Interventions: Procedure: Sham Osteopathic Manipulative Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — The investigators wish to see if emergency medicine physicians can use osteopathic evaluation and OMT to reliably treat headaches. The results of the examination and treatment will be recorded, but will not be used to change treatment or to change additional tests.
  Arms: Osteopathic Manipulative Treatment
Procedure: Sham Osteopathic Manipulative Treatment — The sham group will receive 3 sham treatments.
  Arms: Sham Osteopathic Manipulative Treatment

SUMMARY:
PURPOSE The purpose of this research is to determine whether osteopathic manipulative therapy (OMT) is a useful adjunct in evaluation and treatment of headaches.

PROCEDURES If a practitioner determines that a patient has a significant headache he/she may order tests. He/ She may give the patient medications to treat the headache.

The investigators will also ask permission to evaluate and treat the headache using osteopathic evaluation and Osteopathic Manipulative Treatment (OMT). The bedside evaluation and treatment will be performed by an emergency medicine resident. Osteopathic evaluation and OMT is not standard of care for this condition. The investigators also may call the patient in 7 days to see how they are doing.

The investigators wish to see if emergency medicine physicians can use osteopathic evaluation and OMT to reliably treat headaches. The results of the examination and treatment will be recorded, but will not be used to change treatment or to change additional tests. The investigators wish to see whether in the future they can use OMT in certain cases instead of or in conjunction with medications. The investigators plan on asking 50 patients to participate.

DETAILED DESCRIPTION:
Will the Use of Osteopathic Manipulative Treatments on Patients with Headache in the Emergency Department Result in Decreased Pain on 100 Point Pain Scale? PROTOCOL

Patients will be triaged to the appropriate part of the Emergency Department in the usual fashion. A healthcare provider will evaluate the patient and if the patient's chief complaint is headache the provider will determine if they are a candidate for the study utilizing exclusion criteria for the study TABLE 1.

___ Table 1. Exclusion Criteria for the Study

* Temperature 100.4 or greater
* Healthcare provider suspects meningitis, brain abscess, encephalitis
* Altered mental status
* History of trauma
* Cyclic vomiting
* Abdominal migraines
* Analgesic medication taken prior to treatment within an hour
* Providing physician suspects intracranial hemorrhage
* Focal deficits or other neurological abnormalities that lead providing physician to suspect a pathologic process in which osteopathic treatment would not be safe for the patient
* Providing physician feels osteopathic treatment would not be safe for the patient

If patients have none of the above criteria, they may be selected for the study by the Providing Physician.

The provider will ask the patient to rate their initial pain by drawing a vertical line on the 100 mm visual analog scale (VAS) on the Physician Provider Data Form.

The provider will then alert an osteopathic emergency medicine resident to enroll the patient into the study. The resident will then obtain informed consent from the patient and will then take an envelope containing a piece of paper stating whether the patient is to receive the actual osteopathic treatment or if the patient will receive placebo/sham treatment.

Treatment will be performed by osteopathic emergency medicine residents. Each resident has undergone training in Osteopathic Manipulative Techniques (OMT) in their respective medical schools and has fulfilled the requirements for competency in these techniques for graduation.

The osteopathic treatment group will have performed on them 3 standardized osteopathic manipulative treatments. These treatments are muscle energy to the occipital area; muscle energy to the paraspinal muscles bilaterally and facilitated positional release without axial compression. If at any time the patient is unable to tolerate a treatment secondary to pain that particular study will be stopped. At no time will the patient's medical treatment in the emergency department be delayed to perform OMT.For example, if the patient's nurse enters the room with medication, the study will be stopped and patient will not be included in the study. The sham group will receive 3 sham treatments. The patient consent form and information as to whether or not the patient received osteopathic manipulative treatment will be kept in a locked file. The information will be transferred to a password-protected computer file.

After the standardized treatment or sham treatment is performed, the resident will leave the patient and the providing physician will then ask the patient to draw a vertical line on the VAS to again rate their pain.

The providing physician will then place the data form into the envelope that also contains the information about whether the patient received the osteopathic treatment vs. the sham treatment, without seeing the actual information.

Data will then be analyzed and kept in a password-protected file.

ELIGIBILITY:
Inclusion Criteria:

Patients will be triaged to the appropriate part of the Emergency Department in the usual fashion. A healthcare provider will evaluate the patient and if the patient's chief complaint is headache the provider will determine if they are a candidate for the study utilizing exclusion criteria for the study -

Exclusion Criteria:

Exclusion Criteria for the Study

Temperature 100.4 or greater

Healthcare provider suspects meningitis, brain abscess, encephalitis

Altered mental status

History of trauma

Cyclic vomiting

Abdominal migraines

Analgesic medication taken prior to treatment within an hour

Providing physician suspects intracranial hemorrhage

Focal deficits or other neurological abnormalities that lead providing physician to suspect a pathologic process in which osteopathic treatment would not be safe for the patient

Providing physician feels osteopathic treatment would not be safe for the patient

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Headache Pain as Measured by a VAS | Immediately before and after intervention (less than 30 minutes)
  The primary outcome will be the change in pain before and immediately after intervention as measured by a 100 mm visual analog scale (VAS) for pain in patients with headaches that meet the inclusion criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve McGerald, DO, Principal Investigator — Good Samaritan Hospital Medical Center
Locations (1):
- Good Samaritan Hospital Medical Center, West Islip, New York, United States